CLINICAL TRIAL: NCT02705157
Title: The OPTIMAL Study - A Prospective Cohort of Patients With Bone Metastases of the Long Bones
Acronym: OPTIMAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, PD Sander Dijkstra, MD PhD, MD PhD, Leiden University Medical Center
Other Study IDs: NL54439.058.15
Record Dates: First submitted 2016-02-25; First posted 2016-03-10 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Bone Metastasis
Keywords: long bones; survival; prognosis; treatment; quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bone metastasis of the long bone: Patients with bone metastases of the long bone(s) receiving surgical stabilisation of a pathologic or impending fracture or receiving radiotherapy for a painful metastasis.
  Interventions: Procedure: Stabilisation of (impending) pathological fracture; Radiation: Radiotherapy of bone metastasis

INTERVENTIONS:
Procedure: Stabilisation of (impending) pathological fracture — Stabilisation of pathological fracture or impending fracture with prosthesis, plate, intramedullary nail, cement, or other stabilisation method
Radiation: Radiotherapy of bone metastasis — Radiotherapy of bone metastasis, single or multi-fractionated

SUMMARY:
Rationale: Bone metastases arise in 50% of all patients dying from carcinoma, increasing up to 70% in patients with breast and prostate cancer. The lesions can cause pain and fractures, leading to diminished quality of life and poorer survival. Current knowledge concerning adequate, personalized treatment of metastatic lesions of the long bones in patients with disseminated cancer is insufficient and inconclusive due to lack of large, prospective series with patient reported outcome measures.

Objective: The OPTIMAL cohort aims to describe the quality of life and pain perception of patients after local treatment (radiotherapy and/or surgery) of metastases of the long bones, for both the entire cohort as well as for specific treatments separately. With this a more personalized treatment for metastases in the long bones based on expected survival and impending fracture risk can be provided in order to improve functioning and the quality of life for the remaining lifetime in patients with disseminated cancer.

Study design: Observational, prospective, multicentre cohort study.

Study population: All patients with metastases of the long bones visiting a radiation oncologist or orthopaedic surgeon.

Main study parameters/endpoints: Primary endpoints are patient reported quality of life (including functioning) and pain levels. Complications and survival are secondary endpoints.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients in the OPTIMAL cohort will perhaps not directly benefit from their participation. Participation will contribute to deriving patient-specific treatment modalities for future patients with bone metastases of the long bones. Risks associated with participation in the prospective cohort are considered negligible due to the observational nature of the study. The burden for the patients lies in completion of questionnaires, which is considered to be in proportion with the potential value of this research.

DETAILED DESCRIPTION:
The OPTIMAL Study in its entirety aims to provide a more personalized treatment for metastases in the long bones based on expected survival and impending fracture risk in order to improve functioning and the quality of life for the remaining lifetime in patients with disseminated cancer. The OPTIMAL Study will provide the infrastructure for a prospective cohort (OPTIMAL cohort) and multiple independent trials. The specific aims of the cohort are discussed in this protocol. The objectives and plan of the first trial (Post-Operative Radiotherapy; PORT study) are discussed in a separate protocol.

The primary aim of the cohort is to describe the quality of life and pain perception of patients after local treatment (radiotherapy and/or surgery) of metastases of the long bones, for both the entire cohort as well as for specific treatments separately.

Secondary aims are to describe the complication rate and survival of patients after local treatment (radiotherapy and/or surgery) of metastases of the long bones.

The specific aims of further future individual trials will be described in separate protocols and submitted to the medical research ethics committee (METC) independently. In general however, all trials will be pragmatic research trials in search of answers to which treatment (radiotherapy or surgery) fits specific patients (categorised by metastasis location, expected survival and fracture risk) best.

STUDY DESIGN The cohort will be prospectively collected and multicentre, including all consecutive patients with bone metastases of the long bones (BMLB) who have signed informed consent. These patients will be followed prospectively, and data concerning patient and treatment characteristics as well as patient reported outcomes on quality of life will be collected. Baseline data will be collected by the physician and entered into the OPTIMAL database. These baseline data match the information that is obtained for standard care. For the assessment of patient reported outcomes a set of internationally and nationally validated questionnaires will be used.

At moment of inclusion baseline patient data will be collected for the OPTIMAL cohort, which will also be used for the Post-Operative RadioTherapy (PORT) study. Data will comprehend information concerning demographics, medical history, and clinical status and functioning. Details concerning the treatment(s) will be reported when relevant.

Patients will be invited to fill out questionnaires about quality of life (QoL) at baseline (pre-treatment; if possible), and 4, 8, 12, and 24 weeks after initial treatment, then every six months for minimal two years or until death. All subsequently or concomitantly symptomatic metastases will be registered (including treatment and follow-up), but a new course of questionnaires will generally not be initiated. These outcome measures will be applied in the entire OPTIMAL cohort.

Pain:

Pain has been chosen as primary endpoint because it can act as a proxy for mechanical complications (i.e. loosening). Mechanical complications are only relevant for these patients if they give clinical complaints needing treatment.

To measure the primary endpoint patients will be asked to score the worst pain in the past 24 hours on a numeric rating scale (NRS) from 0-10. In addition, patients will be asked to list their usual pain medication and the escape medication they used the previous 24 hours. These questions are derived from the Brief Pain Intervention (BPI) score, which is advised by the International Consensus Statement for Bone Metastasis Research. The BPI is a pain assessment tool for use with cancer patients developed by the Pain Research Group of the World Health Organization (WHO) Collaborating Centre for Symptom Evaluation in Cancer Care and is also available in Dutch. However, multiple questions are similar to questions in the European Organization for Research and Treatment of Cancer (EORTC) Quality of life questionnaire for palliation (QLQ-PAL15) and EORTC Quality of life questionnaire for bone metastases (QLQBM-22) (described below). Thus to spare patients answering the same questions twice, the investigators have selected only 2 questions from the BPI.

Quality of life:

For longitudinal assessment of quality of life after treatment, the investigators will use nationally and internationally used, validated and recommended questionnaires: European Organization for Research and Treatment of Cancer (EORTC) QLQ-C15-PAL and EORTC QLQ-BM22. In addition, the EQ-5D (5 dimension) questionnaire will be conducted. The EORTC is currently developing a utility scoring instrument for the EORTC QLQ-C30 (from which the QLQ-C15-PAL originates). The investigators expect this scoring instrument will also be applicable for the QLQ-C15-PAL. After validation of this scoring instrument has taken place, the investigators plan to apply it to the data. This would make the addition of the EQ-5D questionnaire redundant and it will then be withdrawn.

Function:

For assessing improvements in functional outcomes after treatment, the Toronto Extremity Salvage Score (TESS) for upper and lower extremities will be used.

Observational clinical data will be collected at baseline (pre-treatment; if possible) and at first, and possibly second, post-operative follow-up (generally, patients are subsequently only seen if there are complications or new complaints):

Complications:

For complication rate, the Henderson classification of complications will be applied. This classification identifies five primary modes of endoprosthetic failure: soft tissue failure (type 1), aseptic loosening (type 2), structural failure (type 3), infection (type 4), and tumour progression (type 5). Wound complications with clinical consequences will be registered separately. Re-operations due to complications will be registered as such in the treatment field as a new operation.

Radiological status:

Progression of BMLB will be monitored with conventional radiography and on indication with CT scan. This is according to usual care, generally at six weeks and 3 months. No additional outpatient visits or imaging will be requested for study purposes only. The radiological images will be used to place the subjective reports of pain (as reported by the patient on a numeric rating scale) into perspective.

Survival:

Dates of death will be derived from the Hospital Electronic Patient Registry, which is linked to the Municipal Personal Records Database. If this is not possible or not up to date, data will be derived from the general practitioner. The utmost will be tried to prevent sending questionnaires to deceased patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Radiographic or histologic proof of metastatic bone disease
* Histologic diagnosis of the primary tumour or - if the diagnosis is unknown - at least adequate diagnostic investigations into the origin of the metastasis (e.g. dissemination imaging, histology, biopsy)
* Bone metastasis deriving from the bones of the extremities

Exclusion Criteria:

* Primary bone tumours (benign and/or malignant)
* No informed consent signed
* Communication with patient is hampered (e.g. language barrier, severe cognitive impairment, dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients visiting the radiation oncologist or the orthopaedic surgeon of participating centres, for possible local treatment of a symptomatic BMLB or impending fracture, will be registered in the OPTIMAL registry. This includes patients with newly diagnosed metastatic bone disease as well as patients undergoing re-treatment of the same lesion or patients who have received previous treatment for other lesions. Preferably patients are included before the start of treatment, but inclusion can also take place during treatment. When patients are already included in the cohort (for treatment of another metastasis), they will not be included a second time when they present with a second lesion of the long bones. This second lesion will be registered under the same patient number.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life before and after treatment as measured by EQ-5D, EORTC BM-22, and EORTC PAL-15. | 4 weeks, 8 weeks, 3 months, 6 months, 12 months, 18 months, 24 months after treatment
  The influence on the quality of life of a treatment will be measured by several patient reported outcome scores (EQ-5D, EORTC BM-22, and EORTC PAL-15) at several time points after treatment. These will be used to calculate the changes shortly and longer after treatment.
Change in pain before and after treatment as measured by an 11-point numeric rating scale (NRS) | 4 weeks, 8 weeks, 3 months, 6 months, 12 months, 18 months, 24 months after treatment
  The influence of a treatment on the pain will be measured by a reported outcome score (NRS) at several time points after treatment. These will be used to calculate the changes shortly and longer after treatment.
Change in function before and after treatment as measured by the Toronto Extremity Salvage Score (TESS). | 4 weeks, 8 weeks, 3 months, 6 months, 12 months, 18 months, 24 months after treatment
  The influence of a treatment on the function will be measured by a patient reported outcome scores (TESS) at several time points after treatment. These will be used to calculate the changes shortly and longer after treatment.

SECONDARY OUTCOMES:
Proportion of participants with overall survival at 6 months | 6 months
Proportion of participants with overall survival at 1 year | 1 year
Proportion of participants with overall survival at 2 years | 2 years
Number of patients with complications as reported by physicians | 8 weeks
  For complication rate, the Henderson classification of complications will be applied. This classification identifies five primary modes of endoprosthetic failure: soft tissue failure (type 1), aseptic loosening (type 2), structural failure (type 3), infection (type 4), and tumour progression (type 5). Wound complications with clinical consequences will be registered separately. Re-operations due to complications will be registered as such in the treatment field as a new operation.
Number of patients with complications as reported by physicians | 6 months
  For complication rate, the Henderson classification of complications will be applied. This classification identifies five primary modes of endoprosthetic failure: soft tissue failure (type 1), aseptic loosening (type 2), structural failure (type 3), infection (type 4), and tumour progression (type 5). Wound complications with clinical consequences will be registered separately. Re-operations due to complications will be registered as such in the treatment field as a new operation.
Number of patients with complications as reported by physicians | 1 year
  For complication rate, the Henderson classification of complications will be applied. This classification identifies five primary modes of endoprosthetic failure: soft tissue failure (type 1), aseptic loosening (type 2), structural failure (type 3), infection (type 4), and tumour progression (type 5). Wound complications with clinical consequences will be registered separately. Re-operations due to complications will be registered as such in the treatment field as a new operation.
Number of patients with complications as reported by physicians | 2 years
  For complication rate, the Henderson classification of complications will be applied. This classification identifies five primary modes of endoprosthetic failure: soft tissue failure (type 1), aseptic loosening (type 2), structural failure (type 3), infection (type 4), and tumour progression (type 5). Wound complications with clinical consequences will be registered separately. Re-operations due to complications will be registered as such in the treatment field as a new operation.

CONTACTS AND LOCATIONS:
Overall Officials: Sander Dijkstra, MD PhD, Principal Investigator — Leiden University Medical Center; Yvette van der Linden, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of OPTIMAL Study — http://www.optimal-study.nl